CLINICAL TRIAL: NCT03683641
Title: Extracorporeal Shockwave Therapy in Insertional Achilles Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2016/427
Record Dates: First submitted 2018-09-04; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Insertional Achilles Tendinopathy
Keywords: Insertional Achilles Tendinopathy; Extracorporeal Shock Wave Therapy; Double-blind Randomized Controlled Trial
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock Wave group (Active Comparator): Applying shock wave to patient's Achilles tendon insertion
  Interventions: Device: Extracorporeal Shock Wave Therapy
- Sham Control group (Sham Comparator): Applying sham shock wave to patient's Achilles tendon insertion
  Interventions: Device: Sham Control group

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — Use ESWT on chronic insertional Achilles tendinopathy
  Arms: Shock Wave group
Device: Sham Control group — Use sham ESWT on chronic insertional Achilles tendinopathy
  Arms: Sham Control group

SUMMARY:
There is still limited number of studies in the literature provides insufficient evidence to support the use of ESWT in the treatment of insertional Achilles tendinopathy and the contribution of a placebo effect to the shock waves was not assessed by previous study. So the investigators conducted a double-blinded randomized-controlled trial at the orthopedic out-patient clinic, Department of Orthopedics, Faculty of Medicine Ramathibodi Hospital between December 2016 and June 2018. Hypothesized that ESWT might be effective on insertional Achilles tendinopathy

DETAILED DESCRIPTION:
Participants aged 18-70 years old who were diagnosed as insertional Achilles tendinopathy by foot and ankle specialists: had symptoms of pain and swelling at Achilles insertion more than 6 months; failed other standard conservative treatments for 3 months, i.e., rest, medication, activity modification, stretching exercise, and heel lift orthosis; be able to complete questionnaires; and willing to participate were enrolled. A computerized block-of-four random numbers were generated into 2 groups; ESWT and placebo (sham) group. Investigators concealed the treatment allocation by sequential sealed opaque envelops. The sealed opaque envelops were opened just before the assigned treatment began. The outcome assessment in this study was seven times at pre-intervention, 2nd, 3rd, 4th, 6th, 12th and 24th weeks. The participants had to complete questionnaire of VAS and VAS-FA Thai version. The investigators used mean and standard deviation for continuous variables, and frequency (%) for categorical data. For non-normally distributed variables, median and range was presented. Continuous data of both interventions was compared using either unpaired t-test or Mann-Whitney U test based on normal distribution. While categorical data was compared using Fisher's exact test. Repeated measures with Bonferroni post hoc analysis was applied for each intervention according to times of follow-up, and between groups. Bartlett's test for equal variances was checked the assumption before using analysis of variance. If the data did not meet the assumption, non-parametric Kruskal-Wallis was performed. The investigators used STATA 15.0 Program, College Station, Texas, USA for all statistical analysis. P-value < 0.05 defined as a significant level. Sample size was estimated using STATA 15.0 Program based on alpha error 0.05, beta error 0.2, mean VAS in controls 5.0, mean VAS in intervention group 3.5, standard deviation (SD) of both group 2.3,(13) pre-intervention assessment for 1 time, post-intervention assessment for 6 times, correlation between the first and the last VAS assessment 0.8. The calculated sample size was 12 per group. With 20% increment for loss of follow-up, the final sample size was 15 per group. All of them remained in the randomized groups and analyzed as intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as insertional Achilles tendinopathy
* Have symptom at least 6 months
* Willing to participate

Exclusion Criteria:

* History of peritendinous steroid injections within 4 weeks
* Neurological conditions
* Local skin infection
* Ankle arthritis, traumatic, inflammation or deformity of ankle
* History of ankle surgery
* Contraindication for ESWT : Hemophilia, Coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Up to 24 weeks
  Visual Analog Scale of Pain on Achilles tendon, range 0-10, 0 means no pain and 10 is the most severe pain

SECONDARY OUTCOMES:
Visual Analog Scale - Foot and Ankle Thai version | Up to 24 weeks
  Range 0-100, 0 is worse, 100 is the best. Having 20 questions. Categorized into Pain, Function and other complaints
The amount of rescue drug use | Up to 24 weeks
  Tablet/day,if amount of drug use is higher mean it is worse
Complications | Up to 52 weeks
  Investigator collected complication such as pain during procedure, tendon rupture, or surgical rate and calculated the NNH